CLINICAL TRIAL: NCT04540614
Title: Upper Cross Syndrome Rehabilitation by Means of Habitual Treatment Plus Strengthening of the Dorsal Erector Muscles. Controlled Clinical Trial.
Brief Title: Upper Cross Syndrome Rehabilitation Strengthening of the Dorsal Erector Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martín, Carlos García (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MartinCG
Record Dates: First submitted 2020-05-22; First posted 2020-09-07 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-02

CONDITIONS: Neck Pain
Keywords: chronic neck pain; upper crossed syndrome; rounded shoulder posture
MeSH Terms: conditions — Neck Pain; Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 70 participants receiving active comparator treatment plus experimental
  Interventions: Other: Strengthening exercises programme
- Control (Active Comparator): 70 participants receiving active comparator treatment
  Interventions: Other: Strengthening exercises programme

INTERVENTIONS:
Other: Strengthening exercises programme — Strengthening exercises for Deep Cervical Flexors, Shoulder external rotators, scapular adductors and thoracic erector muscles

SUMMARY:
The purpose of this study is to determine which treatment is more effective for chronic neck pain associated with Upper Cross Syndrome.

DETAILED DESCRIPTION:
Patients will divided in two groups, control and intervention. Control Group will do exercises of strengthening of Deep Cervical Flexors, Shoulder External Rotators and Adduction of Scapulae.

Intervention group will do the same plus Strengthtening of Erector Thoracic.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain for at least 3 months
* 52º or less in the craniovertebral angle
* 50º or less in the shoulder angle

Exclusion Criteria:

* herniated disk, radiculopathy, diseases of the spine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | 0 week
  tha angle formed by the horizontal line through C7 and the line formed between C7 and the tragus of the ear
Craniovertebral angle | 4 week
  tha angle formed by the horizontal line through C7 and the line formed between C7 and the tragus of the ear
Craniovertebral angle | 8 week
  tha angle formed by the horizontal line through C7 and the line formed between C7 and the tragus of the ear
Shoulder angle | 0 week
  the angle formed by the horizontal line through C7 and the line formed between C7 and the acromion
Shoulder angle | 4 week
  the angle formed by the horizontal line through C7 and the line formed between C7 and the acromion
Shoulder angle | 8 week
  the angle formed by the horizontal line through C7 and the line formed between C7 and the acromion
VAS | 0 week
  The Visual Analogue Scale 0 no pain 10 worst pain
VAS | 4 week
  The Visual Analogue Scale 0 no pain 10 worst pain
VAS | 8 week
  The Visual Analogue Scale 0 no pain 10 worst pain

SECONDARY OUTCOMES:
Muscle Strenght | 0 week
  Muscle strenght tested by a hand held dynamometer
Muscle Strenght | 4 week
  Muscle Strenght tested by a hand held dynamometer
Muscle Strenght | 8 week
  Muscle strenght tested by a and held dynamometer
Muscle Activity | 0 week
  Muscle activity tested by Portable EMG
Muscle Activity | 4 week
  Muscle activity tested by Portable EMG
Muscle Activity | 8 week
  Muscle activity tested by Portable EMG

CONTACTS AND LOCATIONS:
Overall Officials: Carlos García, Principal Investigator — Fisiosesto
Locations (1):
- Fisiosesto, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No